CLINICAL TRIAL: NCT00105963
Title: Parents Helping Infants Study: Preventing Shaken Baby Syndrome and Child Abuse
Brief Title: Prevention of Shaken Baby Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harborview Injury Prevention and Research Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: HIPRCSBS-01
Record Dates: First submitted 2005-03-18; First posted 2005-03-21 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-03

CONDITIONS: Child Abuse; Shaken Baby Syndrome
Keywords: abuse
MeSH Terms: conditions — Shaken Baby Syndrome

INTERVENTIONS:
Behavioral: Education about infant crying

SUMMARY:
This research project seeks to implement an early intervention program that can be effective in the prevention of Shaken Baby Syndrome (SBS) and infant abuse. Our hypothesis is that the Period of PURPLE Crying intervention program can reduce shaking and abuse of infants through changes in knowledge, attitudes and behaviors about early infant crying, especially inconsolable crying. In this 3-year project, we will implement and evaluate an intervention program in selected prenatal classes, hospitals, and primary care pediatric practices.

In this randomized, controlled trial, we will enroll a total of 3000 women/families who are about to give birth or have just given birth to a healthy infant. At each of the three sites (newborn nursery, pediatrician offices and prenatal classes), we will enroll 1000 subjects. Half of all subjects will receive intervention materials (a video, pamphlet and bib/burp cloth) about infant crying. The other half, the control group, will receive comparable materials on infant safety. All subjects will be asked to complete a brief questionnaire at the time of enrollment (pre test), review the materials they receive, complete the Baby's Day Diary for 4 days when the infant is 5 weeks of age and complete a telephone questionnaire (post test) when the infant is 8 weeks of age.

DETAILED DESCRIPTION:
The specific goals of the program are:

1. To change the understanding (i.e., knowledge and attitudes) and reduce the frustration of parents of new infants about the normality of the frustrating properties of crying;
2. To change the behavior of parents to increase caregiving contact in response to crying but to 'walk away' if frustrated;
3. To provide parents with the ability to communicate to other caregivers (relatives, baby-sitters) the knowledge and behavior to reduce frustration induced by inconsolable crying;
4. To provide effective knowledge, skills and teaching materials to health care providers in direct contact with parents concerning crying, shaking and abuse;
5. To reduce the incidence of physical abuse and shaken baby syndrome under one year;
6. To have the Period of PURPLE Crying program adopted as a nationwide early intervention project.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be new parents or parents to be who are either: 1) attending participating prenatal classes; 2) delivering a baby at the participating hospital; or 3) visiting a PSPRN (Puget Sound Pediatric Research Network) pediatrician for infant care.
* Only parents of infants born at > 34 weeks gestation are eligible.

Exclusion Criteria:

* Parents of infants who have serious medical conditions.
* Parents who don't speak and read English.
* Parents of infants born at < 34 weeks gestation.

Ages: 1 Day to 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000
Dates: Start 2005-01; Study Completion 2006-08

PRIMARY OUTCOMES:
Knowledge and attitudes about crying, shaking and abuse
Caregiver behavior
Parenting sense of competence
Maternal depression

CONTACTS AND LOCATIONS:
Locations (1):
- Harborview Injruy Prevention and Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Radesky JS, Zuckerman B, Silverstein M, Rivara FP, Barr M, Taylor JA, Lengua LJ, Barr RG. Inconsolable infant crying and maternal postpartum depressive symptoms. Pediatrics. 2013 Jun;131(6):e1857-64. doi: 10.1542/peds.2012-3316. Epub 2013 May 6. PMID 23650295
- See also: Related Info — http://www.hiprc.org